CLINICAL TRIAL: NCT01652547
Title: A Phase I, Exploratory, Intra-patient Dose Escalation Study to Investigate the Preliminary Safety, Pharmacokinetics, and Anti-tumor Activity of Pasireotide (SOM230) s.c.Followed by Pasireotide LAR in Patients With Metastaticmelanoma or Metastatic Merkel Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230X2404
Record Dates: First submitted 2012-07-12; First posted 2012-07-30 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2016-03

CONDITIONS: Metastatic Melanoma and Merkel Cell Carcinoma
Keywords: Melanoma; Merkel cell carcinoma; Metastatic skin cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Merkel Cell; Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pasireotide sub-cutaneous formulation (Experimental): Pasireotide, will be administered to all patients by s.c. injection, beginning with a dose of 300 μg administered three times daily (t.i.d.) for 2 weeks. If no pasireotide-related clinically meaningful/uncontrolled grade 3 or grade 4 adverse events occur the dose will be administered to all patients at an increased dose of 600 μg t.i.d. for 2 weeks, followed by 2 weeks of 900 μg t.i.d. and followed by 2 weeks of 1200 μg t.i.d. After the 8 weeks period, patients will be kept on treatment drug (highest dose without clinically meaningful/uncontrolled AEs), switched to the corresponding pasireotide LAR dose and followed up for an extra 6 months.
  Interventions: Drug: Pasireotide sub-cutaneous formulation
- Pasireotide long acting release (Experimental): At the start of the follow-up phase patients will be switched to pasireotide LAR administered intramuscularly every 28 days by using the following conversion algorithm so that the steady state PK exposure (Cmax and Ctrough) of pasireotide will be maintained: 300 μg s.c. t.i.d. fi 20mg LAR i.m. q 28 days 600 μg s.c. t.i.d. fi 40 mg LAR i.m. q 28 days 900 μg s.c. t.i.d. fi 60 mg LAR i.m. q 28 days 1200 μg s.c. t.id. fi 80 mg LAR i.m. q 28 days In addition, all patients will keep the treatment with pasireotide s.c. during the first 2 weeks of the LAR phase. The use of s.c. dosing during the initial 2 week period following the first LAR dose provides an appropriate level of medication during the LAR nadir.
  Interventions: Drug: Pasireotide lon acting release formulation

INTERVENTIONS:
Drug: Pasireotide sub-cutaneous formulation — Pasireotide, will be administered to all patients by s.c. injection, beginning with a dose of 300 μg administered three times daily (t.i.d.) for 2 weeks. If no pasireotide-related clinically meaningful/uncontrolled grade 3 or grade 4 adverse events occur the dose will be administered to all patients at an increased dose of 600 μg t.i.d. for 2 weeks, followed by 2 weeks of 900 μg t.i.d. and followed by 2 weeks of 1200 μg t.i.d. After the 8 weeks period, patients will be kept on treatment drug (highest dose without clinically meaningful/uncontrolled AEs) , switched to the corresponding pasireotide LAR dose and followed up for an extra 6 months.
  Arms: Pasireotide sub-cutaneous formulation
Drug: Pasireotide lon acting release formulation — At the start of the follow-up phase patients will be switched to pasireotide LAR administered intramuscularly every 28 days by using the following conversion algorithm so that the steady state PK exposure (Cmax and Ctrough) of pasireotide will be maintained: 300 μg s.c. t.i.d. fi 20mg LAR i.m. q 28 days 600 μg s.c. t.i.d. fi 40 mg LAR i.m. q 28 days 900 μg s.c. t.i.d. fi 60 mg LAR i.m. q 28 days 1200 μg s.c. t.id. fi 80 mg LAR i.m. q 28 days In addition, all patients will keep the treatment with pasireotide s.c. during the first 2 weeks of the LAR phase. The use of s.c. dosing during the initial 2 week period following the first LAR dose provides an appropriate level of medication during the LAR nadir.
  Arms: Pasireotide long acting release

SUMMARY:
This study will evaluate the preliminary safety, pharmacokinetics, and anti-tumor activity of pasireotide s.c. in patients with metastatic melanoma or metastatic Merkel cell carcinoma. The study consists of three phases: screening, intra-patient dose-escalation, and follow-up phases.

In the screening phase patient will be informed of all aspects of the study and sign informed consent forms and then be screened for study eligibility.

During the intra-patient dose escalation phase, 18 patients will be treated with pasireotide s.c. 300 μg t.i.d. for 2 weeks. If there are no unacceptable AEs, defined as drug-related clinically meaningful, uncontrolled grade 3 or any grade 4 toxicities, patients will be dose escalated to 600 μg t.i.d. for 2 more weeks, then 900 μg t.i.d. for 2 weeks and then 1200 μg for 2 weeks provided that there are no unacceptable AEs. Each patient will be in the dose escalation phase for a maximum of 8 weeks.

At end of the intra-patient dose escalation phase, patients will be allowed to switch to 80 mg pasireotide LAR i.m. q 28 d (or a lower dose in case of toxicity) for an additional 6 months or until disease progression, or unacceptable AEs, or patient withdraws consent. In addition, all patients will keep their pasireotide s.c. t.i.d. treatment (same dose as that at the end of the 8-week dose escalation phase) during the first 2 weeks of the LAR follow-up phase, except on the day receiving the first LAR dose because of an anticipated initial burst of drug release.

ELIGIBILITY:
Inclusion criteria:

1. Patients must have histologically or cytologically confirmed unresectable (stage III) and/or metastatic (stage IV) melanoma or unresectable and/or metastatic Merkel cell carcinoma.
2. Melanoma patients should have no mutation in BRAF and NRAS genes
3. Patients should have lesions that can be biopsied, in addition measurable and non-measurable metastatic lesions and at 1 lesion suitable for 18FDG-PET scan or CT/MRI.
4. ECOG Performance Status of 0 or 1
5. Presence of measurable or non-measurable disease according to RECIST 1.0
6. Adequate organ function: adequate bone marrow function (WBC ≥ 2.5 x 109/L, ANC ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, hemoglobin ≥ 9 g/dL); serum creatinine ≤ 1.5 mg/dL or estimated glomerular filtration rate (eGFR) > 40 ml/min/m2; serum lipase ≤ 1.5 ULN

Exclusion criteria:

1. Patient with primary uveal melanoma
2. Patients with symptomatic CNS metastases who are neurologically unstable or requiring increasing doses of steroids to control their CNS disease
3. Patient who have been previously treated with somatostatin analogue or radiolabeled somatostatin analogs or patients with a known hypersensitivity to somatostatin analogs or any component of the pasireotide s.c. and i.m. formulations or their excipients
4. Patients for whom standard treatment is available and indicated due to rapidly progressive or aggressive disease
5. Patients who received more than 3 prior lines of systemic therapy for the treatment of the disease.
6. Patients receiving any anti-neoplastic therapy within the 4 weeks prior to baseline
7. Patients receiving an investigational drug within 1 month prior to baseline
8. Patients who have undergone major surgery/surgical therapy for any cause within 1 month prior to baseline. Patients must have recovered from the treatment and have a stable clinical condition before entering this study
9. Patients who have received prior radiation therapy ≤ 4 weeks, or limited field radiation ≤ 2 weeks, prior to baseline or the side effects of such therapy have not resolved to ≤ grade 1.
10. Patients unwilling to perform repeated biopsies
11. Patients with known gallbladder or bile duct disease, acute or chronic pancreatitis (patients with asymptomatic cholelithiasis and asymptomatic bile duct dilation can be included)
12. Patients with abnormal coagulation (PT or PTT elevated by 30% above normal limits)
13. Patients on continuous anticoagulation therapy. Patients who were on anticoagulant therapy must complete a washout period of at least 10 days prior to baseline and have confirmed normal coagulation parameters before study inclusion
14. Patients who are not biochemically euthyroid
15. Patients with known history of hypothyroidism are eligible if they are on adequate and stable replacement thyroid hormone therapy for at least 3 months prior to baseline
16. Patients with QT-related exclusion criteria
17. Baseline QTcF >450 ms

    * History of syncope or family history of idiopathic sudden death
    * Known history of prolong QT syndrome
    * Sustained or clinically significant cardiac arrhythmias
    * Patients with risk factors for torsades de pointes such as uncorrected hypokalemia, uncorrected hypomagnesemia, clinically relevant cardiac failure (NYHA class III or IV), clinically significant/symptomatic bradycardia or high-grade AV block
    * Concomitant medications known to prolong the QT interval
    * Known concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes mellitus or Parkinson's disease), HIV, liver cirrhosis, uncontrolled hypothyroidism or cardiac failure
    * Patients with unstable angina, sustained ventricular tachycardia, ventricular fibrillation, high grade (NOT advanced!) heart block or history of acute myocardial infarction less than one year prior to baseline
18. Patients with any of the following severe and/or uncontrolled medical conditions:

    * Uncontrolled diabetes as defined by HbA1c > 8% despite adequate therapy
    * Patients with the presence of active or suspected acute or chronic uncontrolled infection or with a history of immunodeficiency, including a positive HIV test result (ELISA and Western blot)
    * Liver disease or history of liver disease such as cirrhosis, decompensated liver disease, or chronic active hepatitis B and C or chronic persistent hepatitis
    * Life-threatening autoimmune and ischemic disorders
19. Patients who have a history of another primary malignancy, with the exception of locally excised non-melanoma skin cancer and carcinoma in situ of uterine cervix. Patients who had no evidence of disease from another primary cancer for 3 or more years are allowed to participate in the study
20. Pregnant or nursing (lactating) women
21. Women of child-bearing potential
22. Patients with baseline ALT or AST > 3 x ULN or baseline total bilirubin > 1.5x ULN
23. Patients with presence of Hepatitis B surface antigen (HbsAg) or presence of Hepatitis C antibody test (anti-HCV)
24. History of, or current alcohol misuse/abuse within the past 12 months prior to visit 1 (baseline)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of patients with AEs, SAEs | Week 8
  Number of patients with AEs (overall and by severity) SAEs according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Number of patients with laboratory abnormalities and changes in laboratory values | Week 8
  Number of patients with laboratory abnormalities according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Number of patients with electrocardiographic abnormalities and changes in electrocardiograms readings | Week 8
  Number of patients with ECG according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Number of patients with vital sign abnormalities and changes in vital signs | Week 8
  Number of patients with vital sign abnormalities according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0

SECONDARY OUTCOMES:
Changes in laboratory values, electrocardiograms readings, and vital signs values at study completion | Baseline, Day 253
Tumor response according to Response Evaluation Criteria in Solid Tumors (RECIST 1.0) as measured by disease control rate ((DCR), (Complete Response (CR), Partial Response (PR), Stable Disease (SD)) | Baseline, Day 57, Day 113, Day 169, Day 225
  Tumor response as measured by DCR defined as the proportion of patients with best overall response of complete response (CR), partial response (PR) or stable response (SR) according to the RECIST Version 1.0 Criteria.
PK parameters for each cycle on Day 1 (Cmax,d1 Tmax,d1, AUC0-2hr,d1), and on day 8 at steady state (Cmin,d8, Cmaxd8, Tmax,d8, Cavg,d8, AUC0-2hr,d8, ARd8) | Day 1, 8, 15, 22, 29, 36, 43, 50, 57, 85, 113, 141, 169, 197 and 225
  Pasireotide plasma concentrations will be summarized by dose and time and PK profile of pasireotide concentration over time will be generated by dose.
Changes from baseline on melanoma response biomarkers (MIA, S100B) overtime and its correlation with each dose | Baseline, Day 8, 15, 22, 29, 36, 43, 50, 57, 113, 169 and 225
  Melanoma response biomarkers (MIA, S100B) will be evaluated in pre- and post-treatment samples on all patients to assess the biochemical response to pasireotide as change from baseline at Day 8, 15, 22, 29, 36, 43, 50, 57, 113, 169 and 225.
Changes from baseline and/or actual levels of potential response and/or secretion biomarkers over time, in repeated tumor and/or blood samples | Baseline, Day 1, 15, 29, 43, 57, 113, 169 and 225
  PD and cellular effect makers in tumor Protein expression levels for different PD markers such as p4EBP-1, pS6, pAKT, pERK and for different cellular effect markers of proliferation and apoptosis (such as Ki67, cyclin D1, cleaved caspase, PARP), angiogenesis (such as microvessel density) and secretion (such as IGF-1 receptor); change from baseline of these markers at day 29 and 57.
Number of patients with AEs, SAEs at study completion | Day 253
  Number of patients with AEs (overall and by severity) SAEs according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0
Number of patients with electrocardiographic abnormalities and changes in electrocardiograms readings at study completion | Day 253
  Number of patients with ECG abnormalities according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Number of patients with laboratory abnormalities and changes in laboratory values at study completion | Day 253
  Number of patients with laboratory abnormalities according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0
Number of patients with vital sign abnormalities and changes in vital signs at study completion | Day 253
  Number of patients with vital sign abnormalities and changes in vital signs according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Novartis Investigative Site, Essen, Germany
- Switzerland (2):
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich

REFERENCES:
- See also: Results for CSOM230X2404 on the Novartis Clinical Trial Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=14789